CLINICAL TRIAL: NCT00474188
Title: A Phase II, Multicenter, Single-Arm, Open-Label Study to Evaluate the Safety and Efficacy of Lenalidomide (Revlimid ®) in Combination With Dexamethasone in Subjects With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study to Evaluate Lenalidomide Combined With Dexamethasone in Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Celgene Corporation (Industry)
Responsible Party: Robert Knight, M.D., Celgene/sponsor
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-NHL-005
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2009-09-02 (Estimated); Status verified 2009-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Celgene; Revlimid; Lenalidomide; Diffuse Large B-cell lymphoma; Non-Hodgkins lymphoma; CC-5013; Response Rate; Tumor Control Rate; Duration of Response; Time to Progression; Progression-free survival and safety
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: CC-5013 (lenalidomide); Drug: dexamethasone

INTERVENTIONS:
Drug: CC-5013 (lenalidomide) — Lenalidomide 25 mg, orally, once daily, on Days 1 to 21 of every 28-day cycle administerd in combination with dexamethasone 40 mg, orally, once daily, on Days 1, 8, 15, and 22 of every 28-day cycle
  Other Names: CC-5013; lenalidomide; Revlimid
Drug: dexamethasone — Dexamethasone 40 mg, orally, once daily, on Days 1, 8, 15, and 22 of every 28-day cycle administered in combination with lenalidomide 25 mg, orally, once daily, on Days 1 to 21 of every 28-day cycle.
  Other Names: Decadron

SUMMARY:
To evaluate the safety and efficacy of lenalidomide (Revlimid ®) in combination with dexamethasone in subjects with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma (NHL) can be divided into two general prognostic groups: the indolent lymphomas and the aggressive lymphomas. Indolent lymphomas have a relatively good prognosis, with median survival time as long as 10 years, but they are not usually curable in advanced stages. Aggressive NHL constitutes about half of all cases of NHL in North America and Western Europe. Of the aggressive lymphomas, diffuse large B-cell lymphoma (DLBCL) is the most common type, accounting for up to 30 percent of newly diagnosed cases. The aggressive type of NHL has a shorter natural history; approximately 50-60% of these subjects can be cured with combination chemotherapy regimens. Even with recent advances, many patients with advanced stage DLBCL are not cured with conventional therapy. This leaves a subset of subjects who will eventually relapse or who are refractory to treatment.

Due to the variation in the clinical behavior of the different types of aggressive NHL, it is important to test lenalidomide in DLBCL. Other studies are addressing the activity of lenalidomide in the other types of aggressive lymphomas, as well as in indolent NHL. It is important to test lenalidomide in combination therapy. This study is focused on treating subjects with relapsed or refractory DLBCL using oral lenalidomide in combination with oral dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diffuse large B-cell non-Hodgkin's lymphoma
* Relapsed or refractory to previous therapy for non-Hodgkin's lymphoma
* Measurable disease on cross sectional imaging that is at least 2 cm in the longest diameter
* ECOG performance score of 0,1 or 2
* Willing to follow the pregnancy precautions

Exclusion Criteria:

* Any of the following laboratory abnormalities.
* Absolute neutrophil count (ANC) < 1,500 cells/mm3 (1.5 x 109/L).
* Platelet count < 60,000/mm3 (60 x 109/L).
* Serum SGOT/AST or SGPT/ALT 5.0 x upper limit of normal (ULN).
* Serum total bilirubin > 2.0 mg/dL (34 µmol/L).
* Subjects who are candidates for and willing to undergo an autologous stem cell transplant.
* History of active CNS lymphoma within the previous 3 months
* Subjects not willing or unable to take DVT prophylaxis
* History of other malignancies within the past year
* Positive HIV or active Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, MD, Principal Investigator — The Alfred
Locations (24):
- United States (19):
  - Palo Verde Hematology/Oncology, Ltd., Glendale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Advanced Medical Specialties, Miami, Florida
  - Hematology/Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington Heights, Illinois
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Southwest Oncology Associates, Lafayette, Louisiana
  - Washington County Hospital, The Center for Clinical Research, Hagerstown, Maryland
  - Kalamazoo Hematology & Oncology, Kalamazoo, Michigan
  - Oncology & Hematology Specialists, PA, Denville, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northwestern Carolina, Oncology and Hematology PA, Hickory, North Carolina
  - New Bern Cancer Care, New Bern, North Carolina
  - James Cancer Hospital, Columbus, Ohio
  - SouthWest Regional Cancer Center, Austin, Texas
  - Northern Utah Associates, Ogden, Utah
- Australia (4):
  - The Alfred Hospital, Melbourne, Victoria
  - Frankston Hospital, Frankston
  - HOCA, South Brisbane
  - Border Medical Oncology, Wodonga
- Cross Cancer Institute, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide in Combination With Dexamethasone: Lenalidomide 25 mg administered orally once daily on Days 1-21 every 28 days, in combination with dexamethasone 40 mg administered orally on Days 1, 8, 15, and 22 of each 28-day cycle.
Period: Overall Study
Arm/Group | Lenalidomide in Combination With Dexamethasone
Started | 26
Completed | 20 (Disease progression=15, adverse event=4, death=1)
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — Study discontinued by sponsor | 5

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 66.7 (11.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Region of Enrollment [Number; unit: participants]
  Australia | 4
  Canada | 2
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate
Description: Number of participants demonstrating complete or partial tumor response (Cheson B, Horning S, Coiffier B, Shipp M, Fisher R, Connors J, et al, Report of an international workshop to standardize response criteria for non-Hodgkins' lymphoma. J Clin Oncol.1999;17:1244-53).
  Study terminated prematurely. Analysis not conducted.
Time Frame: One Year
Population: Study terminated prematurely. Analyses of efficacy not conducted.
Measure: Mean (95% Confidence Interval); unit: Participants
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 0

2. Secondary Outcome: Tumor Control Rate
Description: Number of participants demonstrating complete tumor response, partial tumor response, or stable disease.
  Study terminated prematurely. Analysis not conducted.
Time Frame: One Year
Measure: Mean (95% Confidence Interval); unit: Participants
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response
Description: Time from first demonstration of at least a partial response to the first documentation of disease progression, including death due to non-Hodgkin's lymphoma.
  Study terminated prematurely. Analysis not conducted.
Time Frame: One year
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression
Description: Time from the start of study drug therapy to the first documentation of disease progression.
  Study terminated prematurely. Analysis not conducted.
Time Frame: One year
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: Time from the start of study drug therapy to the first observation of disease progression or death due to any cause.
  Study terminated prematurely. Analysis not conducted.
Time Frame: One year
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Lenalidomide in Combination With Dexamethasone
Number analyzed (Participants) | 0

LIMITATIONS AND CAVEATS:
Study terminated prematurely as a business decision. Analyses of efficacy not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present the data generated from the study provided that the investigator shall (i) furnish the sponsor with a copy of any proposed publication or presentation at least thirty (30) days in advance of the submission of such material, (ii) delete from such material any confidential information of the sponsor, and (iii) delay submission of same for up to sixty (60) days to permit the preparation and filing of intellectual property applications.